CLINICAL TRIAL: NCT02264145
Title: The Effect of Alcoholic-carrier Solutions Within-devices (HFA134a-MDI or Respimat®) on Breath Alcohol Measured by Ethylometer in Healthy Volunteers
Brief Title: The Effect of Alcoholic-carrier Solutions Within Devices (HFA134a-MDI or Respimat®) on Breath Alcohol Measured by Ethylometer in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 260.3171
Record Dates: First submitted 2014-10-14; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (4):
- Ethanolic Solution From HFA134a-MDI - low (Experimental)
  Interventions: Drug: Ethanolic Solution From HFA134a-MDI - low
- Ethanolic Solution From HFA134a-MDI - medium (Experimental)
  Interventions: Drug: Ethanolic Solution From HFA134a-MDI - medium
- Ethanolic Solution From HFA134a-MDI - high (Experimental)
  Interventions: Drug: Ethanolic Solution From HFA134a-MDI - high
- Ethanolic Solution From Respimat® (Experimental)
  Interventions: Drug: Ethanolic Solution From Respimat®

INTERVENTIONS:
Drug: Ethanolic Solution From HFA134a-MDI - low
  Arms: Ethanolic Solution From HFA134a-MDI - low
Drug: Ethanolic Solution From HFA134a-MDI - medium
  Arms: Ethanolic Solution From HFA134a-MDI - medium
Drug: Ethanolic Solution From HFA134a-MDI - high
  Arms: Ethanolic Solution From HFA134a-MDI - high
Drug: Ethanolic Solution From Respimat®
  Arms: Ethanolic Solution From Respimat®

SUMMARY:
The study objective is to determine the effect of the ethanolic solutions inhaled from the Metered dose inhaler (MDI) (15.5 mg, 31.2 mg and 62.4 mg of ethanol) and from Respimat® (18.4 of ethanol) on the breath alcohol measurements in healthy volunteers.

Secondary aim is to determine the linear dose-effect for the HFA 134a-MDI doses. An open, randomized, four-way-cross-over design is chosen. The randomization is balanced and stratified in accordance with predicted values of the volunteers of Total Lung Capacity (TLC)

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoker volunteers without dental prothesis
* 18 to 45 years old, male or female
* No clinically significant abnormal conditions at the screening visit. A clinically significant disease is defined as one, which in the opinion of the investigator, may either put the subject at risk because of participation in the study, or a disease which may influence the results of the study or the subjects ability to participate in the study
* Volunteer with gamma-glutamyl-transferase (GGT) level < 32 IU/L
* Volunteer is able to sign informed consent in accordance with Good Clinical Practice and local legislation
* Volunteers is able to be trained in the performance of technically satisfactory pulmonary function tests
* Volunteer is able to be trained in the correct use HFA-MDI, Respimat® and Ethylometer
* Affiliated to the National Social Security System

Exclusion Criteria:

* Subjects who are already taking other investigational drugs or who have taken part in another trial during the past month
* Consumption of alcoholic beverage within 12 hours prior to observation period
* Breast feeding or pregnant female or female with no medically approved contraception method (oral contraceptive, intra uterine device)
* Subjects who have a known intolerance or hypersensitivity to aerosolized containing products and/or to any of the HFA-MDI or Respimat® excipient
* Volunteer with history of drug abuse and/or alcoholism
* Intensive exercise one week prior to the study
* Major exposure to dust, smoke or pollution one week prior to the study
* Subjects with an upper or lower respiratory tract infection within the previous four weeks to screening. This is to insure no reduced alcohol absorption by mucus
* Current psychiatric disorders
* Previous inclusion in the randomized period of this study
* Subjects on concomitant medications

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 1998-11; Primary Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) of blood alcohol level estimated from breath alcohol concentration after the four formulation inhalations | up to 15 min after inhalation

SECONDARY OUTCOMES:
Breath alcohol concentration profile within each formulation | up to 15 min after inhalation
Maximum duration of alcohol detection exhaled air (Td) for each formulation | up to 15 min after inhalation
Highest breath alcohol concentration measured (Cmax) | up to 15 min after inhalation
Time to highest breath concentration (Tmax) | up to 15 min after inhalation
Number of patients with adverse events | up to 5 days